CLINICAL TRIAL: NCT06658925
Title: The Safety and Efficacy of Olverembatinib as Maintenance Therapy or Preemptive Therapy After Allo-HSCT in Adult Ph + Acute Lymphoblastic Leukemia
Brief Title: Olverembatinib as Maintenance Therapy or Preemptive Therapy After Allo-HSCT in Ph+ALL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024065
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Ph+ Acute Lymphoblastic Leukemia (Ph+ALL); HSCT; Tyrosine Kinase Inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olverembatinib as maintenance therapy or preemptive therapy post-HSCT (Experimental): Olverembatinib is used to prevent recurrence or preemptive treatment after transplantation.
  Interventions: Drug: Olverembatinib is used to prevent recurrence or preemptive treatment after transplantation.

INTERVENTIONS:
Drug: Olverembatinib is used to prevent recurrence or preemptive treatment after transplantation. — Olverembatinib is used to prevent recurrence or preemptive treatment after transplantation.

SUMMARY:
This study is a single-center, prospective, single-arm exploratory study. Ph + acute lymphoblastic leukemia patients treated with allogeneic hematopoietic stem cell transplantation were recruited from the Stem Cell Transplantation Center of the Hospital of Hematology, Chinese Academy of Medical Sciences. The number of patients is expected to be 50 cases. The enrolled patients plan to receive Olverembatinib as a post-transplant treatment regimen, including maintenance therapy to prevent recurrence and preemptive treatment. Hematopoietic reconstitution ( neutrophil > 0.5 × 10 ^ 9 / L, platelet > 50 × 10 ^ 9 / L ) was evaluated after enrollment. From 2 months to 3 months after transplantation, Olverembatinib 40 mg QOD was added for maintenance treatment until 2 years after transplantation. During maintenance treatment, Olverembatinib dose ( dose range 20 mg QOD to 40 mg QOD ) can be adjusted according to blood picture, biochemical index or other oral drugs ( triazole drugs, etc. ).

ELIGIBILITY:
Inclusion Criteria:

* ( 1 ) Acute lymphoblastic leukemia with positive Ph chromosome or BCR / ABL fusion gene ; after allogeneic hematopoietic stem cell transplantation, and survived for more than 30 days after transplantation.

( 2 ) Age older than or equal to 18 years old ( 3 ) Informed consent can be signed by themselves. ( 4 ) Adequate organ function must be met : renal function and liver function are as follows : serum creatinine is 2 times lower than the normal upper limit, AST, ALT and ALP are lower than the normal upper limit of 3 times, and total bilirubin is lower than the normal upper limit of 3 times ( if the liver GVHD is clearly diagnosed, less than or equal to 5 × ULN ) ).

( 5 ) HIV negative, HBV and HCV negative. ( 6 ) The Eastern Oncology Collaborative Group Physical Status Assessment ( ECOG-PS ) was 0-2 points.

( 7 ) Informed consent must be signed before the start of the study procedure, and the informed consent must be signed by the patient himself or his immediate family. Considering the patient 's condition, if the patient 's signature is not conducive to the treatment of the disease, the informed consent is signed by the legal guardian or the patient 's immediate family.

Exclusion Criteria:

* ( 1 ) Hematology remission was evaluated at 1 month after transplantation, and complete donor chimerism was achieved.

( 2 ) Severe cardiovascular diseases ( including myocardial infarction, unstable angina pectoris, severe arrhythmia and congestive heart failure, etc. ) occurred during the previous use of the third generations of TKI treatment.

( 3 ) Uncontrolled infection at the time of enrollment ; severe complications of mechanical ventilation or hemodynamic instability ; those who had undergone autologous or allogeneic stem cell transplantation; ( 4 ) The serological reaction of known HIV or active hepatitis C virus is positive ; ( 5 ) suffering from mental illness or other illness and can not cooperate with the research treatment and monitoring requirements ; ( 6 ) being unable or unwilling to sign the consent ; ( 7 ) pregnant or lactating women ; ( 8 ) Patients with other special conditions who were assessed as unqualified by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
2-year RFS after transplantation | 2 year after HSCT
  2-year relapse-free survival after transplantation